CLINICAL TRIAL: NCT02103257
Title: Sequential Icotinib Plus Chemotherapy Versus Icotinib Alone as First-line Treatment in Stage IIIB/IV Lung Adenocarcinoma: a Randomized, Open-label, Multicenter Study
Brief Title: Sequential Icotinib Plus Chemotherapy Versus Icotinib Alone as First-line Treatment in Stage IIIB/IV Lung Adenocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV62
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Drug Therapy; Pemetrexed; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential icotinib plus chemotherapy (Experimental): Sequential icotinib plus chemotherapy : pemetrexed 500mg/m2 iv d1, cisplatin 75mg/m2 d1, icotinib 125 mg is administered orally three times per day d 8-21, every 3 weeks for a cycle. After receiving a maximum of 4 cycles treatment, non-progressive patients continue to receive icotinib as maintenance treatment until disease progression or intolerable toxicity.
  Interventions: Drug: Sequential Icotinib Plus Chemotherapy
- Icotinib (Active Comparator): Icotinib 125 mg is administered orally three times per day until disease progression or intolerable toxicity.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Sequential Icotinib Plus Chemotherapy — Sequential icotinib plus chemotherapy: pemetrexed 500mg/m2 iv d1, cisplatin 75mg/m2 d1, icotinib 125 mg is administered orally three times per day d 8-21, every 3 weeks for a cycle. After receiving a maximum of 4 cycles treatment, non-progressive patients continue to receive icotinib as maintenance treatment until disease progression or intolerable toxicity.
  Other Names: ALIMTA; DDP; Comana, BPI-2009
  Arms: Sequential icotinib plus chemotherapy
Drug: Icotinib — Icotinib 125 mg is administered orally three times per day until disease progression or intolerable toxicity.
  Other Names: Comana; BPI-2009
  Arms: Icotinib

SUMMARY:
This randomised, controlled, multicentre trial is designed to assess the efficacy and safety of sequential icotinib plus chemotherapy versus single icotinib as first-line treatment in stage IIIB/IV lung adenocarcinoma patients with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of lung adenocarcinoma with measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded on CT)
* Patients must have previously untreated locally advanced or metastatic NSCLC
* EGFR activating mutation (exon 19 deletion, L858R) is required
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1

Exclusion Criteria:

* Prior chemotherapy or treatment with gefitinib, erlotinib, or other drugs that target EGFR
* Patients with wild-type EGFR
* Any other investigational agents are not permitted
* Any evidence of interstitial lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 15 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.
Objective response rate | 15 months
  Number of subjects with confirmed objective response according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Adverse events | 24 months
  The number of patients who suffered adverse events, which is graded by NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, MD, Principal Investigator — Tang-Du Hospital
Locations (31):
- China (31):
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou military region general hospital, Lanzhou, Gansu
  - General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Cancer Hospital of Sun Yat-sen, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Jiangmen central hospital, Jiangmen, Guangdong
  - The university of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Medical Oncology,Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Thoracic Surgery,Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Guangdong Agribusiness Center Hospital, Zhanjiang, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan Provincal Nong Ken Hospital, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Medical Oncology，General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Radiation Oncology，General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Respiratory medicine，General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Baoji Central Hospital, Baoji, Shanxi
  - 3201 Hospital, Hanzhong, Shanxi, Hanzhong, Shanxi
  - Shaanxi province people's hospital, Xi’an, Shanxi
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Chang'an Hospital, Xi’an, Shanxi
  - Tangdu Hospital，Fourth Military Medical University, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Cancer Hospital, Xi’an, Shanxi
  - Urumqi General Hospital of Lanzhou Military Region General Hospital, Ürümqi, Xinjiang
  - Xinjiang medical university affiliated tumor hospital, Ürümqi, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Autonome Region Xinjiang Uygur Chinese medicine hospital, Ürümqi, Xinjiang